CLINICAL TRIAL: NCT01084369
Title: Phase IV: Effect of Testosterone on Endothelial Function and Microcirculation in Type 2 Diabetic Patients With Hypogonadism
Brief Title: Effect of Testosterone on Endothelial Function and Microcirculation in Type 2 Diabetic Patients With Hypogonadism
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Withdrawal of sponsorship
Sponsor: Tameside Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Edward Jude, Consultant Physician, Tameside Hospital NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Testosterone version1
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Type 2 Diabetes; Hypogonadism
Keywords: Type 2 diabetes; Hypogonadism; Testosterone; Endothelial dysfunction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypogonadism | interventions — Testosterone; testosterone undecanoate; Vardenafil Dihydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Testosterone, Vardenafil (Experimental): All patients will receive Testosterone (n=40) of these (10 patients) will also receive Vardenafil
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Testosterone — NEBIDO ampoules containing a solution for injection of 1000mg/4ml of testosterone undecanoate. NEBIDO injection 1000mg/4ml will be given at baseline, 6 weeks, 18 weeks, 30 weeks, 42 and 54 weeks. Levitra will be given to those patients with erectile dysfunction for 2 weeks in addition to Nebido.
  Concomitant medication deemed necessary by the investigator as part of the routine clinical management will be permissable.
  Other Names: Testosterone (NEBIDO); Vardenafil (Levitra)

SUMMARY:
Diabetes mellitus is associated with long-term complications affecting mainly the eyes, nerves and kidneys. One of the main underlying causes for this is damage to the lining of the small blood vessels supplying these organs with dysfunction of the endothelium (lining of the small blood vessels). Testosterone has been shown to have an effect macro (large) blood vessels with limited data available on the micro (small) blood vessels. Testosterone is recognised to have important effects on metabolism and vascular behaviour beyond the accepted effects on secondary sexual characteristics. Physiological testosterone therapy is associated with some beneficial effects on the cardiovascular system and has been used with some success to treat patients with stable angina and chronic heart failure. The investigators therefore propose to study the effects of testosterone replacement therapy in patients with hypogonadism (low testosterone levels) on the endothelium in males with type 2 diabetes. 40 diabetic patients with type 2 diabetes and low testosterone levels and erectile dysfunction (impotence) will be recruited into the study. All patients will receive testosterone replacement therapy and 10 patients will also receive Vardenafil (a drug used to treat impotence). The investigators hope to demonstrate an improvement in endothelial dysfunction by assessing biochemical markers such as nitric oxide (a chemical that causes relaxation for the blood vessels) and C-reactive protein (a chemical that can increase in patients with diabetes) as well as the effect on weight, blood pressure, diabetes control and cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* 40 male patients with type 2 diabetes mellitus.
* T2DM as judged by WHO criteria:

  * onset of diabetes mellitus after the age of 30 years
  * blood glucose controlled by diet or drugs other than insulin, or insulin initiated after 2 years diagnosis of diabetes
  * no history of diabetic ketoacidosis.
* Symptomatic Hypogonadism as defined by:

  * Total testosterone below 10 nmol/l
  * Aging males' symptom score (AMS) above 36.
* Hypogonadic men with erectile dysfunction
* Age range- 50-80 years

Exclusion Criteria:

* Patients with uncontrolled hypertension (BP>145/95 on treatment) or significant hypotension. (BP<100 systolic)
* Current smokers
* Recent myocardial infarction (<6 months), unstable angina or ongoing chest pain, recent (within 6 months) cardiac intervention (e.g. angioplasty, stenting or CABG) or stroke.
* Patients with clinical nephropathy (24 hr protein >0.5 g or urine protein +) or moderate renal failure (serum creatinine >150 micromol/l).
* History of prostate cancer or suspicion of prostate cancer on clinical examination
* Androgen dependent carcinoma of the male mammary gland
* Liver tumours
* Hypersensitivity to NEBIDO or LEVITRA
* Polycythaemia
* General systemic illness, including cardiac, renal or hepatic insufficiency
* Patients on nitrates will not be included in the Levitra arm.
* History of loss of vision in one eye because of non arteritic ischaemic optic neuropathy (NAION), regardless of whether this episode was in connection or not with previous PDE5 inhibitor exposure.
* Hereditary degenerative retinal disorders such as retinitis pigmentosa.
* Clinically significant chronic haematological disease which may lead to priapism
* Bleeding disorders
* Significant active peptic ulceration.
* Concomitant use of vardenafil with HIV protease inhibitors such as ritonavir and indinavir is contraindicated, as they are potent inhibitors of CYP 3A4
* Concomitant use of vardenafil with potent CYP 3A4 inhibitors ketoconazole and itraconazole (oral form) is contra-indicated in men older than 75 years.
* Patients deemed unable to comply with the requirements of the protocol.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-10-11 (Actual); Primary Completion 2014-09-14 (Actual); Study Completion 2014-09-14 (Actual)

PRIMARY OUTCOMES:
Improvement in endothelial dependent and endothelial-independent vasodilatation | 30 and 54 weeks
  Improvement in markers of endothelial function

SECONDARY OUTCOMES:
Markers of endothelial function | 54 weeks
  Secondary efficacy variables will include changes of the following
  * Availability of nitric oxide
  * Endothelial inflammation as measured by CRP
  * Serum levels of endothelial markers: IGF and adhesion molecules
  * BMI, waist circumference, glycaemic control (HbA1c), lipid profile and blood pressure.
  * Other laboratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Edward Jude, MD, MRCP, Principal Investigator — Tameside Hospital NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Tameside General Hospital, Ashton-under-Lyne, Lancashire
  - Tameside Hospital NHS Foundatoin Trust, Ashton-under-Lyne